CLINICAL TRIAL: NCT06160999
Title: TABRIE: Trusted Faces, Familiar Places (CGHE)
Brief Title: Improving Uptake of Pediatric Vaccines Through Religious Conferences and Vaccines-in-a-van in Aceh, Indonesia
Acronym: TABRIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Abram Wagner, Assistant Professor of Epidemiology and Research Assistant Professor, Global Public Health, School of Public Health, University of Michigan
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00235620
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Vaccination

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge design with a cross-sectional sampling structure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Religious Conference (Experimental): Clusters will have religious conference.
  Interventions: Behavioral: Religious conferences
- Religious Conference control (No Intervention): Clusters will have not religious conference. Clusters' background characteristics matched to the Conference arm.
- Vaccine-in-a-van (Experimental): Clusters will have deployment of a mobile vaccine clinic ("vaccine-in-a-van").
  Interventions: Behavioral: Vaccine-in-a-van
- Vaccine-in-a-van control (No Intervention): Clusters will not have a deployment of a mobile vaccine clinic ("vaccine-in-a-van"). Clusters' background characteristics matched to the Van arm.

INTERVENTIONS:
Behavioral: Religious conferences — The conference will invite local subdistrict-level imams and other religious leaders, along with a range of community health workers, including those not traditionally trained to give vaccines. During the conference there will be some sessions with everyone, and some that are broken down by profession. The conference topics will be developed in conjunction with the religious leaders, but will focus on the importance of infant health
  Arms: Religious Conference
Behavioral: Vaccine-in-a-van — For the vaccine-in-a-van concept, our community health worker will travel to different areas in the test subdistricts. These locations will be decided on in conjunction with the local health department and the research team's knowledge of the area. We will target areas which would have families with young children, particularly: schools, mosques, and sports fields. The purpose of the van will be to bring vaccines to the community, but also to put a human face (our community health worker) to vaccines outside of a clinical setting.
  Arms: Vaccine-in-a-van

SUMMARY:
The goal of this cluster, randomized controlled trial is to study the impact of mobile vaccine clinics and religious conferences on pediatric vaccination coverage. The main questions will be: does vaccination coverage change in geographic areas with the mobile vaccine clinics vs those areas without mobile vaccine clinics; and does vaccination coverage change in geographic areas with religious conferences on vaccination vs those areas without religious conferences. In repeated surveys, adult participants will respond about their children's vaccination status. Participants will not be individually randomized to the interventions. Rather, their geographical area will be randomized.

DETAILED DESCRIPTION:
This project seeks to create a paradigm shift in how the public views and utilizes vaccination services. Currently, community health centers remain the default setting for vaccination, and clinicians the default administrators. However, the general population may have difficulty accessing these clinics or trusting traditional vaccination providers, particularly if they are members of marginalized communities that have experienced medical discrimination. This project applies a two-pronged approach by addressing issues of trust and ease of access among the general population. This project is innovative by: a) mobilizing religious communities to discuss vaccines (to counter reported lack of information about vaccines among unvaccinated families) and b) training more community health workers in vaccination and in physically delivering vaccines through a "Vaccine-in-a-van" concept to facilitate ease in accessing vaccines. By mobilizing these individuals in the community settings where people live, work, worship, and learn, this project will expand vaccine information and services.

More specifically, this project plans to work with local health leaders in a low vaccination community in Aceh, Indonesia to identify social institutions that are part of children and families' daily lives; these could include houses of worship, schools, or community centers. This project will fund a mobile vaccine delivery unit to go to these locations to physically bring vaccines to the people and to link them with existing immunization clinic infrastructure. This project will also work towards changing the culture of child health and vaccination through substantial discussions and conversations with multiple levels of religious leaders at conferences.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18+, and
* Proficient in Bahasa Indonesia, and
* Plan to live in neighborhood for next year
* Parent of child <5, or
* Planning to have a child within next year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Full vaccination | Records from vaccination cards or clinic records 6 months since the start of the intervention
  Number of participants fully vaccinated. Full vaccination means 1 dose of BCG; 3 doses of DTP; 3 doses of polio vaccine; 1 dose of measles-containing vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Abram Wagner, PhD, Principal Investigator — University of Michigan
Locations (1):
- Universitas Syiah Kuala, Banda Aceh, Special Region of Aceh, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Reproducibility and replicability of studies are both extremely important. Therefore, we plan to upload a final dataset (along with code detailing my statistical analysis) to a public repository. This dataset will have personally identifiable information removed - and the geographic location will be coded by a number to prevent individuals being able to locate members of the study and identify them.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Study data will be made available by December 31, 2026
Access Criteria: This will be publicly available.

REFERENCES:
- [Derived] Ladhania R, Ichsan I, Koumpias AM, Yufika A, Indah R, Liansyah TM, Wagner AL, Harapan H. Improving uptake of pediatric vaccines through religious conferences and mobile vaccine clinics in Aceh, Indonesia (TABRIE): study protocol for a stepped wedge cluster randomized controlled trial. Trials. 2025 Nov 21;26(1):528. doi: 10.1186/s13063-025-09170-5. PMID 41272880